CLINICAL TRIAL: NCT02505685
Title: Dynamic PET CT as a Tool for Treatment Efficacy Monitoring in Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Nir Peled, Professor, Rabin Medical Center
Other Study IDs: 0618-14-RMC
Record Dates: First submitted 2015-07-02; First posted 2015-07-22 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-10

CONDITIONS: Lung Cancer
Keywords: Lung; Cancer; Biomarkers; PET-CT; Early detection
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung cancer: People that were diagnosed with advanced lung cancer.

SUMMARY:
The purpose of this study is to evaluate the use of Dynamic PET/CT as a tool to assess disease response to anti-cancer therapy in Lung Cancer patients.

DETAILED DESCRIPTION:
Background:

Lung cancer is a devastating disease in which the response for first line therapy is only 30%. Evaluating response is performed normally by a CT or PET-CT scans after 2-3 cycles of therapy, thus, lack of response is been evaluated only after the patient has been treated following significant amount of therapy, which is inefficient in 70% of cases.

Therefore, there is an urgent need to develop tools that might predict response to therapy during the early course of therapy; Most valuable will be before or after the first cycle of therapy. For that reason, the investigators aim in this study to evaluate the use of Dynamic PET-CT as a tool to assess disease response to anti-cancer therapy in Lung Cancer patients.

Objectives:

1. To assess the feasibility of baseline Dynamic PET-CT as a tool for assessing response for anti-cancer therapy in Lung Cancer patients.
2. To predict early response to treatment as soon as after 1 cycle of therapy by dynamic and static PET-CT.
3. To correlate Dynamic PET-CT with survival/disease free survival

Method:

200 advanced lung cancer patients will be enrolled over 3 years in a single institute, single arm study at Rabin Medical Center, Beilinson Hospital.

Patients will be evaluated by a Dynamic PET-CT protocol: before initiation of therapy, 7-14 days after the first therapy cycle, 3 months after initiation of therapy and 6 months after the first therapy cycle. In addition, non-invasive biomarkers that are routinely measured including protein markers (CEA- Carcinoembryonic Antigen, CYFRA21- Cytokeratin 19 Fragment, NSE- Neuron Specific Enolase) will be assessed in this trial.

Disease response will be evaluated by Response Evaluation Criteria In Solid Tumors (RECIST criteria).

Additional PET-CT will not increase radiation dose significantly. The mean estimated radiation dose for a limited CT of the chest is about 14 mSv (i.e., 7mSv for limited diagnostic CT and FDG ([18F]-fluorodeoxyglucose), each). The dynamic stage will add radiation dose of about 0.3mSv. Of note, the significance of adding radiation dose is less of importance with regard to treatment of patients with aggressive cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Lung cancer, stage 4
* Patients are planned to be treated by a systemic anti-cancer therapy.
* A define lesion for imaging.
* Able and willing to sign an informed consent form.
* First line therapy or at least 6 weeks after previous line of therapy

Exclusion Criteria:

* Pregnant or lactating women.
* Anti cancer therapy within the last 6 weeks before enrollment.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced lung cancer patients (Stage 4)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Compare baseline PET-CT with PET-CT after 7-14 days. | 12 months

SECONDARY OUTCOMES:
Evaluate disease-free survival (DFS) in lung cancer by using dynamic PET-CT. | 12 months
Evaluate overall survival rate (OS) in lung cancer by using dynamic PET-CT. | 12 months
Measuring response to treatment by PET-CT. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nir Peled, MD PhD FCCP, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No
article will be released